CLINICAL TRIAL: NCT01787162
Title: Screening for Pulmonary Vascular Changes in Patients With Chronic Myeloproliferative Diseases
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 24-393 ex 11/12
Record Dates: First submitted 2012-10-10; First posted 2013-02-08 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Myeloproliferative Disorders; Pulmonary Hypertension
Keywords: Myeloproliferative disorders; pulmonary hypertension; pulmonary vascular diseases
MeSH Terms: conditions — Myeloproliferative Disorders; Hypertension, Pulmonary | interventions — Cardiac Catheterization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples with DNA will be retained for later examinations at the Biobank, in case that the patient agrees (extra patient information).
  The blood samples are taken only during routine tests.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- myeloproliferative disorders: Echocardiography, spiroergometry, cardiac catheterization
  Interventions: Other: Echocardiography, spiroergometry, cardiac catheterization

INTERVENTIONS:
Other: Echocardiography, spiroergometry, cardiac catheterization — patients with CMPD will undergo echocardiography, spiroergometry, and right heart catheterization, if indicated

SUMMARY:
Goal of the study is to assess the frequency of pulmonary hypertension in patients with chronic myeloproliferative diseases. In each patient an echocardiography at rest will be performed. In patients without musculoskeletal disease an exercise test (spiroergometry) will be performed. Patients with elevated SPAP at rest or with reduced exercise capacity (peak VO2 < 65%) a right heart catheterization (RHC) will be recommended. Also patients with advanced NYHA functional class (III or IV) or with typical PH findings in electrocardiogram will be advised to undergo a RHC. Additionally for the evaluation of exercise capacity a 6 MWD will be performed.

This work- up of patients allows clinical and hemodynamic evaluation.

DETAILED DESCRIPTION:
Previous small studies and clinical cases have suggested a possible association between pulmonary hypertension (PH) and chronic myeloproliferative disorders (CMPD). MPD may cause PH through different mechanisms as: high cardiac output, asplenia, direct obstruction of pulmonary arteries by megakaryocytes, chronic thromboembolic endothelial pulmonary hypertension (CTEPH), porto-pulmonary hypertension (POPH). However, the exact prevalence of PH in this group of disorders is not known.

This study is designed to identify the pulmonary vascular changes and describe the prevalence of pulmonary hypertension (defined in this study as mean pulmonary arterial hypertension (mPAP) ≥25mmHg as assessed by right-heart catheterization (RHC) or systolic pulmonary arterial pressure (sPAP) ≥37mmHg (2.9 m/s) assessed by echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Patients with myeloproliferative disorders
* Written informed consent

Exclusion Criteria:

* Manifest pulmonary hypertension
* Significant pulmonary disease
* Left-sided heart failure or diastolic compliance dysfunction
* Hemodynamic relevant valvular disease
* Systemic arterial hypertension (at rest systolic >150 mmHg, diastolic > 90 mmHg, during exercise > 220 mmHg)
* Severe anemia
* Uncontrolled supraventricular and ventricular arrhythmias
* Myocardial infarction (within the last 12 months)
* Pulmonary embolism (within the last 12 months)
* Recent therapy changes (within the last 12 months)
* Recent major surgeries (within the last 12 months)
* For exercise tests: musculoskeletal diseases which may unable the exercise tests

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with myeloproliferative disorders
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2012-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
pulmonary arterial pressure | at baseline

SECONDARY OUTCOMES:
change of pulmonary arterial pressure | between baseline and after 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Horst Olschewski, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Pulmonology, Graz, Austria